CLINICAL TRIAL: NCT02142179
Title: Impact of a Curriculum Intervention on Asthma Knowledge in Adolescents of a Public School in Salvador-Bahia-Brazil
Acronym: KARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado da Bahia (Other)
Responsible Party: Principal Investigator, Ana Carla Carvalho Coelho, NP, Msc, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KARE-001
Record Dates: First submitted 2014-05-11; First posted 2014-05-20 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Asthma
Keywords: Asthma; Knowledge; School-Based Service; Adolescents
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KARE Intervention (Experimental): KARE - Knowledge about Asthma and Respiratory Education is an educational curriculum intervention organized with school staff to be applied to the intervention group. This intervention will consist of theoretical - practical weekly workshops with a targeted content for asthma and involves aspects related to anatomy and physiology of the respiratory tract, conceptualization of asthma, prevention, treatment, maintenance and retrieval; recognition and actions in periods of exacerbations and use the action plan. These workshops are suitable for the course plan of disciplines sciences, biology, chemistry, physics, history, geography, portuguese and mathematics. Those are characterized as a mandatory curriculum component and they should be developed for all students.
  Interventions: Behavioral: Knowledge about Asthma and Respiratory Education (KARE)
- A traditional curriculum education. (No Intervention): The control group will receive a traditional curriculum education.

INTERVENTIONS:
Behavioral: Knowledge about Asthma and Respiratory Education (KARE) — KARE - Knowledge about Asthma and Respiratory Education is an educational curriculum intervention organized with school staff to be applied to the intervention group. This intervention will consist of theoretical - practical weekly workshops with a targeted content for asthma and involves aspects related to anatomy and physiology of the respiratory tract, conceptualization of asthma, prevention, treatment, maintenance and retrieval; recognition and actions in periods of exacerbations and use the action plan. These workshops are suitable for the course plan of disciplines sciences, biology, chemistry, physics, history, geography, portuguese and mathematics. Those are characterized as a mandatory curriculum component and they should be developed for all students.
  Arms: KARE Intervention

SUMMARY:
The purpose of this study is to estimate the impact of a curriculum intervention on asthma knowledge in adolescents of a public school in Salvador-Bahia-Brazil.

DETAILED DESCRIPTION:
Asthma is one of major causes of morbidity and mortality due to chronic diseases worldwide with higher mortality and morbidity in adolescents. Interventions directed to adolescents and systematically developed within the school environment has been performed around the world. In spite of that, studies such Bruzzese (2004; 2011) have already shown that clinical interventions associated with educational activities in group composed of individuals with similar lifestyles and characteristics are able to modify the behavior of the individual as well as reduce emergency room visits and hospitalizations. Thus, it is necessary to develop this study.

This study is a controlled clinical trial. The intervention will be a curriculum intervention on asthma. This intervention will consist of theoretical - practical weekly workshops with a targeted content for asthma and involves aspects related to anatomy and physiology of the respiratory tract, conceptualization of asthma, prevention, treatment, maintenance and retrieval; recognition and actions in periods of exacerbations and use the action plan. These workshops are suitable for the course plan of disciplines sciences, biology, chemistry, physics, history , geography, portuguese and mathematics . Those are characterized as a mandatory curriculum component and they should be developed for all students in elementary and secondary education.

In parallel curriculum intervention, the investigators will identify the frequency of individuals with diagnosis/symptoms suggestive of asthma by applying the ISAAC questionnaire and verification of Forced Expiratory Volume in one second (FEV1) using the portable Vitalograph copd - 6. This assessment will identify students with suspected asthma, symptoms suggestive of asthma and asthma diagnosed.

The curriculum will be organized educational intervention with school staff to be applied to the intervention group (it includes all students from 10 to 19 years previously registered. The afternoon shift is defined as the intervention group and may participate asthmatic and non-asthmatic students). It is noteworthy that, subsequently, the same intervention will be performed with the control group (in which students participate in the morning shift and may participate in asthmatic and non-asthmatic students). The intervention group will receive a complementary intervention where questions directed reinforce attitudes in periods of exacerbation and use the action plan, while the control group will receive this same intervention after the study.

The study will be held at the College Presidente Emilio Garrastazu Medici (Currently its name is College Estadual do Stiep Carlos Marighella) which is a school unit with medium-sized and offers all series of the second segment of the Elementary School, Middle School and Professional Education. This school was chosen because of system of evaluation and teaching methodology as well defined in its political pedagogical project.

The investigators will identify the frequency of individuals with diagnosis/symptoms suggestive of asthma by applying the ISAAC questionnaire and verification of Forced Expiratory Volume in one second (FEV1) will monitor all individuals duly registered and allocated in the age group 10-19 years are enrolled in the 5th to 8th grades in this study.

A despite about data Collection Instrument, will be used: 1. Questionnaires ISAAC - International Study of Asthma and Allergies in Childhood; 2. Form to characterize the subjects and clinical outcomes and 3. Structured questionnaires for assessing knowledge (two different data collection instruments):

1. Questionnaires ISAAC - International Study of Asthma and Allergies in Childhood:

   In the first phase of the study, standardized questionnaires developed by ISAAC will be applied. It aims to evaluate symptoms suggestive of asthma. The first part of the questionnaire consists of 8 questions which mainly use 3 questions to estimate the prevalence of asthma : 1 - " Did you ever in your life you (or your child ) had wheezing (wheezing )? " , 2 - "In the last twelve months you (or your child ) had wheezing ( wheezing )?" 3 - "Have you ( or your child ) had asthma?".
2. Form to characterize the subjects and clinical outcomes:

   This form is composed of two parts: the first part consists of demographic and socio biological data and the second parts of issues related to clinical outcomes. The variables are emergency due to asthma in the past year, emergency due to asthma in past 30 days, emergency due to asthma past two weeks, prior oral intubation, hospitalization due to asthma in the last year, ICU admissions, nocturnal awakenings in the last year, nocturnal awakenings in the last 30 days, nighttime awakenings in the last two weeks, daytime last year awakenings, daytime awakenings in the last 30 days, daytime awakenings in the last two weeks, number of days missed at school in the last year, number of days missed at school last month, number of lost subjects (if already deprecated) in the last year, use of control medications, spirometric values. This form must be applied before and after implementation of the intervention.
3. Form for assessing knowledge:

To assess knowledge about asthma and the exacerbation due to this disease, a structured questionnaire that contains 20 questions with three possible answers to all questions will be used: "Yes", "no" and " I do not know". This questionnaire is organized so that a number of questions covering a field but it is not built for the explicit subject in the research.

The areas are: knowledge of the pathology, triggers, treatment, management of crisis and myths/truths so that the researcher can analyze the performance counting the overall score and domains.The adjustments represent the knowledge level of the respondent. Up to 25 % of hits - Poor knowledge; 26 - 50% correct - satisfactory knowledge; 51-75 % accuracy - Good knowledge; 76-100 % correct - excellent knowledge.

Knowledge about learning about relief treatment and maintenance will be carried out through a questionnaire consists of 4 situations that mimic reality. It trys to observe the therapeutic knowledge of the individual in situations of imminent asthma attack , with the following options answer: "never", "rarely", "sometimes" , "often" ,"always".

The investigators will collect data and analyzed in the period from October 2011 to December 2014. Tools of data collection described above and after signing the Informed Consent and the Coordinator of School and after approval of the research by the Ethics Committee - Universidade Federal da Bahia. This protocol was submitted and approved.

The investigators will use the Statistical Programme Statistic Program for Social Sciences (SPSS) version 21.0 to process data. We will analyse data by descriptive statistics (proportions and measures of central tendency), Relative risk (RR) , absolute risk (AR) , odds ratios (OR) and logistic regression analysis to identify the measures of association will be used effect of systematic educational interventions independent of confounding variables. In all analyzes will be considered the significance level of 5 % .

The ethical aspects shall be based on Resolution 196/96 governing research involving human subjects, the resolution 466/2012 and the Code of Ethics for Professional Nursing. The research will respect the basic principles of bioethics: autonomy, non - maleficence, beneficence, and justice, and should be appropriate to scientific principles, rely on free and informed consent of the research subject and / or his legal representative, establish procedures to ensure confidentiality and privacy of the people involved indirectly. The Program will receive the return of the results obtained through research.

ELIGIBILITY:
Inclusion Criteria:

* All students aged 10-19 years enrolled in the College Presidente Emilio Garrastazu Medici (Currently its name is College Estadual do Stiep Carlos Marighella) whose present the Statement of Consent Form signed by parents/ tutors and by themselves;
* Individuals of the same age with symptoms suggestive of asthma and/or previous diagnosis as well as those without asthma after signing the Statement of Consent Form may be included;

Exclusion Criteria:

* Individuals not willing to participate of the study;
* Individuals who have not signed the consent form;
* Individuals with cognitive impairment and with any special needs must not be included in this study.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 181 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Knowledge about asthma in adolescents of a public school in Salvador-Bahia- Brazil at 3 months | Baseline; up to 2 weeks; up to 3 months; up to 1 year after intervention

SECONDARY OUTCOMES:
Visits to emergency in the subgroup of patients with asthma/ symptoms suggestive of asthma | Baseline; up to 2 weeks and up to 3 months
Hospitalization in the subgroup of patients with asthma/ symptoms suggestive of asthma. | Baseline; up to 2 weeks and up to 3 months
Daytime and nighttime awakenings in the subgroup of patients with asthma/ symptoms suggestive of asthma | Baseline; up to 2 weeks and up to 3 months
Rescue medication use in the subgroup of patients with asthma/ symptoms suggestive of asthma | Baseline; up to 2 weeks and up to 3 months
Use of the action plan in the subgroup of patients with asthma/ symptoms suggestive of asthma | Baseline; up to 2 weeks and up to 3 months
Absenteeism to school in the subgroup of patients with asthma/ symptoms suggestive of asthma | Baseline; up to 2 weeks and up 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Adelmir Souza-Machado, PHD, Study Director — Federal University of Bahia
Locations (1):
- Universidade Federal da Bahia and College Estadual Presidente Emílio Garrastazu Médici (Currently its name is College Estadual do Stiep Carlos Marighella), Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Bruzzese JM, Sheares BJ, Vincent EJ, Du Y, Sadeghi H, Levison MJ, Mellins RB, Evans D. Effects of a school-based intervention for urban adolescents with asthma. A controlled trial. Am J Respir Crit Care Med. 2011 Apr 15;183(8):998-1006. doi: 10.1164/rccm.201003-0429OC. Epub 2010 Dec 7. PMID 21139088
- [Background] Sole D, Wandalsen GF, Camelo-Nunes IC, Naspitz CK; ISAAC - Brazilian Group. Prevalence of symptoms of asthma, rhinitis, and atopic eczema among Brazilian children and adolescents identified by the International Study of Asthma and Allergies in Childhood (ISAAC) - Phase 3. J Pediatr (Rio J). 2006 Sep-Oct;82(5):341-6. doi: 10.2223/JPED.1521. Epub 2006 Aug 28. PMID 16951799
- [Background] Bruzzese JM, Bonner S, Vincent EJ, Sheares BJ, Mellins RB, Levison MJ, Wiesemann S, Du Y, Zimmerman BJ, Evans D. Asthma education: the adolescent experience. Patient Educ Couns. 2004 Dec;55(3):396-406. doi: 10.1016/j.pec.2003.04.009. PMID 15582346
- [Background] Joseph CL, Peterson E, Havstad S, Johnson CC, Hoerauf S, Stringer S, Gibson-Scipio W, Ownby DR, Elston-Lafata J, Pallonen U, Strecher V; Asthma in Adolescents Research Team. A web-based, tailored asthma management program for urban African-American high school students. Am J Respir Crit Care Med. 2007 May 1;175(9):888-95. doi: 10.1164/rccm.200608-1244OC. Epub 2007 Feb 8. PMID 17290041
- [Background] Sole D, Camelo-Nunes IC, Wandalsen GF, Mallozi MC, Naspitz CK; Brazilian ISAAC's Group. Is the prevalence of asthma and related symptoms among Brazilian children related to socioeconomic status? J Asthma. 2008 Jan-Feb;45(1):19-25. doi: 10.1080/02770900701496056. PMID 18259991
- [Background] Akinbami LJ, Schoendorf KC. Trends in childhood asthma: prevalence, health care utilization, and mortality. Pediatrics. 2002 Aug;110(2 Pt 1):315-22. doi: 10.1542/peds.110.2.315. PMID 12165584
- [Background] Bateman ED, Hurd SS, Barnes PJ, Bousquet J, Drazen JM, FitzGerald JM, Gibson P, Ohta K, O'Byrne P, Pedersen SE, Pizzichini E, Sullivan SD, Wenzel SE, Zar HJ. Global strategy for asthma management and prevention: GINA executive summary. Eur Respir J. 2008 Jan;31(1):143-78. doi: 10.1183/09031936.00138707. PMID 18166595
- See also: Global Initiative for Asthma (GINA) — http://www.ginasthma.org